CLINICAL TRIAL: NCT07100015
Title: The Effect of Shoulder Massage and Therapeutic Touch on Pain and Anxiety After Laparoscopic Cholecystectomy: A Three-Arm Single-Blind Randomized Controlled Trial
Brief Title: The Effect of Shoulder Massage and Therapeutic Touch on Pain and Anxiety After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SBFGU
Record Dates: First submitted 2025-06-14; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Massage Therapy; Pain; Anxiety; Theropathic Touch
Keywords: Pain; anxiety,; laparoscopic cholecystectomy,; massage,; theropathic touch
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups; Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): in which patients did not receive any treatment and received routine postoperative care in the clinic.
  Interventions: Device: Control Group
- Therapeutic touch (Experimental): in which therapeutic touch was applied
  Interventions: Device: therapeutic touch
- Shoulder massage group (Experimental): in which shoulder massage was applied
  Interventions: Device: Shoulder massage

INTERVENTIONS:
Device: Control Group — in which patients did not receive any treatment and received routine postoperative care in the clinic
  Arms: Control Group
Device: therapeutic touch — Therapeutic touch applications
  Arms: Therapeutic touch
Device: Shoulder massage — shoulder massage was applied
  Arms: Shoulder massage group

SUMMARY:
This randomized controlled trial compared the effects of shoulder massage and therapeutic touch on pain and anxiety after laparoscopic cholecystectomy. Both interventions significantly reduced pain and anxiety levels compared to the control group. Shoulder massage was more effective in reducing pain, while therapeutic touch was more effective in reducing anxiety. These methods are recommended for broader use in clinical practice.

DETAILED DESCRIPTION:
Background: Laparoscopic cholecystectomy (LC) is a frequently preferred surgical method for treating gallstones. Non-pharmacologic approaches have an important place in addition to pharmacologic treatment methods. Methods such as massage and therapeutic touch are included in the literature as effective alternatives to reduce pain and anxiety.

Aim: This study aimed to compare the effects of shoulder massage and therapeutic touch on shoulder pain and anxiety after laparoscopic cholecystectomy.

Methods: The study was a three-arm randomized controlled trial. After baseline assessment, participants were randomly assigned to three groups; random assignment was done using the Microsoft Excel 2016 program. Participants were divided into three groups: Group 1 (n=24), in which shoulder massage was applied, Group 2 (n=25), in which therapeutic touch was used, and Group 3 (n=25) in which patients did not receive any treatment and received routine postoperative care in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Participants were expected to be able to speak Turkish and have normal verbal communication skills.
* They were required to possess normal cognitive abilities and have no psychiatric diagnoses.
* Patients aged between 18 and 70 years.
* Patients undergoing general anesthesia.
* Patients who voluntarily agree to participate in the research

Exclusion Criteria:

* Patients receiving epidural analgesia post-surgery.
* Patients whose laparoscopic cholecystectomy (LC) procedure was converted to an open cholecystectomy during the operation.
* Patients experiencing postoperative confusion, requiring intensive care, or developing secondary complications that impair their ability to respond to questions accurately.
* Patients who do not report shoulder pain following surgery.
* Patients in a catabolic state, those aged 70 years or older, individuals with chronic pain or opioid use, and those experiencing severe postoperative symptoms such as excessive nausea, vomiting, bleeding, or infection.
* Patients with surgical drains (e.g., Hemovac) may negatively influence pain levels and sleep quality, thereby interfering with the effectiveness of the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
For shoulder pain: Measured with the Visual Analog Scale (VAS). | four month
  Shoulder Pain Intensity Assessed by Visual Analog Scale (VAS)
For anxiety: The State-Trait Anxiety Inventory (STAI) was used. | four month
  State-Trait Anxiety Inventory (STAI) Score for Anxiety Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun Universitesi, Giresun, Piraziz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided